CLINICAL TRIAL: NCT03113760
Title: Multicenter, Double-blind, Placebo-controlled, Randomized Withdrawal Trial With Tadekinig Alfa (r-hIL-18BP) in Patients With IL-18 Driven Monogenic Autoinflammatory Conditions: NLRC4 Mutation and XIAP Deficiency
Brief Title: Therapeutic Use of Tadekinig Alfa in NLRC4 Mutation and XIAP Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AB2 Bio Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NLRC4/XIAP.2016.001
Record Dates: First submitted 2017-02-28; First posted 2017-04-14 (Actual); Results first posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: NLRC4-MAS; XIAP Deficiency
MeSH Terms: conditions — Lymphoproliferative Syndrome, X-Linked, 2 | interventions — interleukin-18 binding protein; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Initial phase of 18 weeks is a single arm, open-label (SAOL) period where Tadekinig alfa is administered in addition to the standard of care treatment used for the control of flares. The SAOL period will be followed by an up to 16-week randomized withdrawal phase (RW). All patients who showed response to treatment at the end of the SAOL phase will be enrolled in the RW phase. In the RW phase patients will be randomized to either Tadekinig alfa or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tadekinig alfa (Experimental): Patients that showed response to treatment in the SAOL phase will receive Tadekinig alfa for up to 16 weeks.
  Interventions: Drug: Tadekinig alfa
- 0.9% sodium chloride (Placebo Comparator): Patients that showed response to treatment in the SAOL phase will receive placebo comparator for up to 16 weeks.
  Interventions: Other: 0.9% sodium chloride

INTERVENTIONS:
Drug: Tadekinig alfa — Tadekinig alfa is a soluble glycoprotein of 164 amino acids produced from Chinese Hamster Ovary cell line. Tadekinig alfa is supplied as a colorless to slightly yellow, sterile solution for injection in glass vials containing sodium chloride, and 0.02M sodium phosphate buffer as excipients. It is available in a concentration of 20mg/0.5mL.
  Other Names: IL-18BP; r-hIL-18BP
  Arms: Tadekinig alfa
Other: 0.9% sodium chloride — To ensure that the treatment remains blinded for the entire study period, the placebo solutions will be supplied in identical vials and similar labelling as the active drug and will be indistinguishable in terms of their texture, color, and smell.
  Arms: 0.9% sodium chloride

SUMMARY:
This is a Phase 3 study to assess the safety and efficacy of Tadekinig alfa in patients with monogenic, interleukin-18 (IL 18) driven autoinflammation due to Nucleotide-binding oligomerization domain, leucine-rich repeat and caspase recruiting domain (CARD domain) containing 4 (NLRC4) - Macrophage activation syndrome (MAS) mutation (NLRC4-MAS mutation) or X-linked inhibitor of apoptosis (XIAP) deficiency. Because of the likelihood for pathogenic IL-18 in certain monogenic diseases, patients known to harbor deleterious mutations in NLRC4-MAS or XIAP and who have a history of ongoing inflammation will be enrolled if they have ferritin ≥ 500 ng/mL or persistent C reactive protein (CRP) elevation ≥ 2 times the upper limit of normal (ULN) and the patients should have a Modified Autoinflammatory Disease Activity Index (mAIDAI) ≥ 4.

DETAILED DESCRIPTION:
The study is designed with single-arm, open-label phase (SAOL) of Tadekinig alfa treatment duration for 18-week followed by an up to 16-week Randomized Withdrawal (RW) period for efficacy and safety evaluation, with no interruption between the two phases of treatment. The screening period will occur before the SAOL phase and before the first dose of Investigational Medicinal Product (IMP)

ELIGIBILITY:
INCLUSION CRITERIA

1. Patients with genetic diagnosis of NLRC4-MAS mutation or XIAP deficiency (caused by BIRC4 gene mutation) as confirmed by analysis performed at the central genetics laboratory. If possible, flow cytometry assay will be performed in parallel to confirm diagnosis of XIAP deficiency. (Note: Previous flow cytometry assay results will be permitted for confirmation of XIAP deficiency diagnosis.)
2. Patients with XIAP deficiency and a previous bone marrow transplantation are allowed, if they show evidence of primary or secondary graft failure, or failure to achieve phenotypic correction with evidence of XIAP-related disease recurrence or clinically significant mixed chimerism.
3. Ferritin ≥ 500 ng/mL or persistent elevation of CRP ≥ 2x ULN and mAIDAI ≥4
4. Patients receiving corticosteroids, non-steroidal anti-inflammatory drugs (NSAIDs) or disease modifying anti-rheumatic drugs (DMARDs), and/or IL-1 blockade with insufficient response to treatment upon enrollment are allowed into the study. Patients not receiving any of these treatments before start of therapy are also allowed.
5. Women of childbearing potential with negative urine pregnancy test (UPT) at all visits (if UPT is positive, a blood test for human chorionic gonadotropin (hCG) to be performed) and who agree to follow highly effective birth control recommendations during the study and until 1 month after the end of the treatment. Birth control methods considered highly effective are: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner or sexual abstinence. In each case of delayed menstrual period (over one month between menstruations, confirmation of absence of pregnancy is strongly recommended. This recommendation also applies to women of childbearing potential with infrequent or irregular menstrual cycles. A post-study contraception duration of 4 weeks is recommended taking into account the median half-life of Tadekinig alfa of almost 40h and 5 half-lives representing a duration of 200 hours.

EXCLUSION CRITERIA

1. Patients with life-threatening co-morbidities not associated with the underlying NLRC4-mutation or XIAP deficiency
2. Positive test for or prior history of HIV, Hepatitis B or Hepatitis C (serology)
3. Presence of active infections or a history of pulmonary TB infection with or without documented adequate therapy
4. Presence of life threatening infections
5. Oncologic causes of symptoms; current or previous history of malignancy
6. Presence of CNS manifestations (i.e. seizures, altered mental status, signs of increased intracranial pressure, chronic papilledema, loss of vision, other sensorineural deficiencies, etc.)
7. Patients suffering from biallelic mutations in any of the following genes: PRF1/Perforin, UNC13D/Munc 13-4, STX11/Syntaxin11, STXB2/Munc 18-2, RAB27A/Rab27a (Griscelli syndrome type 2), LYST (Chediak-Higashi syndrome), AP3B1, ADTB3A, HPS2 mutations (Hermansky-Pudlak syndrome 2) and X-linked lymphoproliferative syndrome (XLP)-1 with SH2D1A mutation
8. Patients who are pregnant or nursing, women of childbearing potential who are unwilling to use highly effective birth control methods (see definition in Inclusion Criteria above) through 4 weeks after the end of their participation in the study
9. Concomitant use of immunosuppression therapies excluded by the protocol. Note: NSAIDs, glucocorticoids, cyclosporine, tacrolimus, and IL-1 inhibitors (anakinra, canakinumab, or rilonacept, or others) are allowed
10. Patients and/or parents (or legal representative, if applicable) not willing to sign assent/informed consent
11. Hypersensitivity to the active substance or one of the excipients of the investigational product

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ed M Behrens, MD, Principal Investigator — Children Hospital of Philadelphia
Locations (9):
- United States (6):
  - UCSD _ Department of Pediatrics / Rady Children's Hospital, La Jolla, California
  - Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital _ Baylor College of Medicine, Houston, Texas
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Providence
- Universitätsklinikum Freiburg, Centrum für Chronische Immundefizienz (CCI) - Paediatric Unit, Freiburg im Breisgau, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
This information will be provided soon

REFERENCES:
- [Derived] Krei JM, Moller HJ, Larsen JB. The role of interleukin-18 in the diagnosis and monitoring of hemophagocytic lymphohistiocytosis/macrophage activation syndrome - a systematic review. Clin Exp Immunol. 2021 Feb;203(2):174-182. doi: 10.1111/cei.13543. Epub 2020 Nov 23. PMID 33128796
- See also: Sponsor details — http://www.ab2bio.com/en/home.8.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm Open-Label - Tadekinig Alfa: The Single Arm Open-Label Full Analysis Set (SAOL-FAS) includes all patients treated with Tadekinig alfa in the first 18 weeks of treatment.
- Randomized Double-Blind Placebo-Controlled - Placebo Arm: The Randomized Double-Blind Placebo-Controlled (RDBPC) Analysis Set includes 1 patient treated with Placebo in the first treatment phase under the initial protocol design starting with a randomized treatment phase. As defined in the study protocol and statistical analysis plan, this patient is excluded from the efficacy analysis due to the difference in treatment schedule but included in the safety analysis.
- Randomized Withdrawal - Tadekinig Alfa Arm: The Tadekinig alfa - Randomized Withdrawal Full Analysis Set (RW-FAS) includes all patients who met the criteria for randomization and were randomized to blinded treatment with Tadekinig alfa in the up to 16 weeks randomized withdrawal phase, which follows the SAOL phase.
- Randomized Withdrawal - Placebo Arm: The Placebo - Randomized Withdrawal Full Analysis Set (RW-FAS) includes all patients who met the criteria for randomization and were randomized to blinded treatment with Placebo in the up to 16 weeks randomized withdrawal phase, which follows the SAOL phase.
Period: Initial 18 Weeks Treatment Phase
Arm/Group | Single Arm Open-Label - Tadekinig Alfa | Randomized Double-Blind Placebo-Controlled - Placebo Arm | Randomized Withdrawal - Tadekinig Alfa Arm | Randomized Withdrawal - Placebo Arm
Started | 14 | 1 | 0 | 0
Completed | 10 | 0 | 0 | 0
Not Completed | 4 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Disease relapse | 1 | 1 | 0 | 0
Period: Randomized Withdrawal Phase
Arm/Group | Single Arm Open-Label - Tadekinig Alfa | Randomized Double-Blind Placebo-Controlled - Placebo Arm | Randomized Withdrawal - Tadekinig Alfa Arm | Randomized Withdrawal - Placebo Arm
Started | 0 | 0 | 5 | 5
Completed | 0 | 0 | 5 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Randomized Double-Blind Placebo-Controlled - Placebo Arm: The Randomized Double-Blind Placebo-Controlled Analysis Set (RDBPC-AS) includes 1 patient treated with Placebo in the first treatment phase.
- Total: Total of all reporting groups
Arm/Group | Single Arm Open-Label - Tadekinig Alfa | Randomized Double-Blind Placebo-Controlled - Placebo Arm | Total
Number analyzed (Participants) | 14 | 1 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 1 | 15
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 10 | 1 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 7 | 1 | 8
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 2 | 1 | 3
  United States | 11 | 0 | 11
  Germany | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Prevention of Flares
Description: The primary outcome measure is the time to first occurrence of disease reactivation during the 16-week RW phase.
  Method of assessment: Biomarkers (CRP / Ferritin) and clinical manifestations of systemic inflammation and end-organ damage.
Time Frame: 16 weeks
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Randomized Withdrawal - Placebo Arm | Randomized Withdrawal - Tadekinig Alfa Arm
Number analyzed (Participants) | 5 | 5
Weeks | 2.71 [1.86 to NA] — Median time to first occurrence of DR was 2.71 weeks for the placebo group and not applicable in the Tadekinig alfa group due to the small number of patients with a disease reactivation. | NA [NA to NA] — Median time to first occurrence of DR was 2.71 weeks for the placebo group and not applicable in the Tadekinig alfa group due to the small number of patients with a disease reactivation.

2. Secondary Outcome: Best Response
Description: Best response to therapy during the SAOL phase including either complete response, partial response or disease improvement.
  Method of assessment: Biomarkers (CRP / Ferritin) and clinical manifestations of systemic inflammation and end-organ damage.
Time Frame: 18 weeks
Population: The safety and efficacy analyses during the SAOL phase is based on the SAOL-FAS as defined in the study protocol and statistical analysis plan. 1 patient treated with Placebo in the first treatment phase under the initial protocol design starting with a randomized treatment phase is excluded from the efficacy analysis due to the difference in treatment schedule but included in the safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Open-Label - Tadekinig Alfa
Number analyzed (Participants) | 14
Participants
  Complete response | 1
  Partial response | 10
  Disease improvement | 3
  No response | 0

3. Secondary Outcome: Duration of Response During the SAOL Phase (Until End of Phase or Disease Reactivation)
Description: Duration of response to therapy during the SAOL phase is assessed for patients having achieved a complete or partial response to therapy during the SAOL phase. It is defined as the time from first evaluation of partial or complete response until the time of subsequent disease reactivation or end of SAOL phase, whichever occurs first.
  Of the 11 patients achieving partial or complete response during the SAOL phase, 8 maintained treatment response until the end of the SAOL phase.
  2 of the 11 patients had a temporary disease reactivation during the protocol mandated steroid weaning in the SAOL phase; 1 of the 11 patients was withdrawn from blinded treatment following a disease reactivation.
Time Frame: The actual mean treatment duration in the SAOL phase was 17.6 weeks (minimum / maximum 5.9 / 22.1 weeks).
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Weeks
Groups:
- Single Arm Open-Label - Tadekinig Alfa - With a Complete or Partial Response to Therapy: Including all patients treated with Tadekinig alfa in the first treatment phase and achieving a complete or partial response to therapy
Arm/Group | Single Arm Open-Label - Tadekinig Alfa - With a Complete or Partial Response to Therapy
Number analyzed (Participants) | 11
Weeks | 11.9 [6.4 to 17.0]

4. Secondary Outcome: Change From Baseline in mAIDAI Total Score in the SAOL Phase
Description: The mAIDAI (modified autoinflammatory disease activitiy index) is an assessment of global disease activity that measures 14 different components for disease as either absent (0 points) or present (2 points for Uveitis 3+/4+ and 1 point for all other symptoms) at each visit. The mAIDAI total score is the sum of the points assigned across all components and ranges from 0 to 15, with a higher score indicating more severe disease activity.
Time Frame: 18 weeks
Population: Change from Baseline to Week 18 in mAIDAI Total Score. The safety and efficacy analyses during the SAOL phase is based on the SAOL-FAS as defined in the study protocol and statistical analysis plan. 1 patient treated with Placebo in the first treatment phase under the initial protocol design starting with a randomized treatment phase is excluded from the efficacy analysis due to the difference in treatment schedule but included in the safety analysis.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Single Arm Open-Label - Tadekinig Alfa
Number analyzed (Participants) | 14
score | -3.9 (0.74)

5. Secondary Outcome: Change From Baseline in Serum Ferritin
Description: Laboratory measure
Time Frame: 34 weeks
Population: Values indicate change from Baseline to End of Phase results. The safety and efficacy analyses during the SAOL phase is based on the SAOL-FAS as defined in the study protocol and statistical analysis plan. 1 patient treated with Placebo in the first treatment phase under the initial protocol design starting with a randomized treatment phase is excluded from the efficacy analysis due to the difference in treatment schedule but included in the safety analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Single Arm Open-Label - Tadekinig Alfa | Randomized Withdrawal - Tadekinig Alfa Arm | Randomized Withdrawal - Placebo Arm
Number analyzed (Participants) | 14 | 5 | 5
ng/mL | -8558.7 (15700.51) | -109.5 (167.4) | 211.8 (359.1)

6. Secondary Outcome: Change From Baseline in Serum CRP
Description: Laboratory measure
Time Frame: 34 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Single Arm Open-Label - Tadekinig Alfa | Randomized Withdrawal - Tadekinig Alfa Arm | Randomized Withdrawal - Placebo Arm
Number analyzed (Participants) | 14 | 5 | 5
ug/mL | -2.28 (4.28) | -0.02 (0.19) | 0.24 (1.35)

7. Secondary Outcome: Resolution of Fevers, Hepato/Splenomegaly and Skin Rash
Description: Clinical assessments if present at Baseline; number displays percentage of patients with resolution of individual disease component at Week 18 or early termination visit based on the number of patients with a baseline assessment for the component of interest.
Time Frame: 18 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of patients with resolution
Arm/Group | Single Arm Open-Label - Tadekinig Alfa
Number analyzed (Participants) | 14
Percentage of patients with resolution
  Resolution of Fever | 100
  Resolution of Organomegaly | 54
  Resolution of Skin rash | 75

8. Secondary Outcome: Improvement in Laboratory Markers - AST (SGOT)
Description: Change from Baseline mean value to Week 18 mean value
Time Frame: 18 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Single Arm Open-Label - Tadekinig Alfa
Number analyzed (Participants) | 14
U/L | -286.2 (727.5)

9. Secondary Outcome: Improvement in Laboratory Markers - ALT (SGPT)
Description: Change from Baseline mean value to Week 18 mean value
Time Frame: 18 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Single Arm Open-Label - Tadekinig Alfa
Number analyzed (Participants) | 14
U/L | -581.2 (1324.21)

10. Secondary Outcome: Improvement in Laboratory Markers - Albumin
Description: Change from Baseline mean value to Week 18 mean value
Time Frame: 18 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Single Arm Open-Label - Tadekinig Alfa
Number analyzed (Participants) | 14
g/L | 4.7 (5.66)

11. Secondary Outcome: Improvement in Laboratory Markers - Hemoglobin
Description: Change from Baseline mean value to Week 18 mean value
Time Frame: 18 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Single Arm Open-Label - Tadekinig Alfa
Number analyzed (Participants) | 14
g/L | 17.2 (18.24)

12. Secondary Outcome: Improvement in Laboratory Markers - Platelets
Description: Change from Baseline mean value to Week 18 mean value
Time Frame: 18 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cells x 10^9/L
Arm/Group | Single Arm Open-Label - Tadekinig Alfa
Number analyzed (Participants) | 14
cells x 10^9/L | 24.0 (143.10)

13. Secondary Outcome: Improvement in Laboratory Markers - Erythrocyte Sedimentation Rate
Description: Change from Baseline mean value to Week 18 mean value
Time Frame: 18 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | Single Arm Open-Label - Tadekinig Alfa
Number analyzed (Participants) | 14
mm/h | -6.3 (10.47)

14. Secondary Outcome: Improvement in Laboratory Markers - Fibrinogen
Description: Change from Baseline mean value to Week 18 mean value
Time Frame: 18 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Single Arm Open-Label - Tadekinig Alfa
Number analyzed (Participants) | 14
mg/dL | 12.7 (108.10)

15. Secondary Outcome: Improvement in Laboratory Markers - D-Dimer
Description: Change from Baseline mean value to Week 18 mean value
Time Frame: 18 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Single Arm Open-Label - Tadekinig Alfa
Number analyzed (Participants) | 14
mg/L | -3.85 (5.89)

16. Secondary Outcome: Hospital Length of Stay
Description: Length of hospitalisation; emergency room attendance and unscheduled visits for treatment of disease reactivations not included
Time Frame: 34 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Single Arm Open-Label - Tadekinig Alfa | Randomized Withdrawal - Tadekinig Alfa Arm | Randomized Withdrawal - Placebo Arm
Number analyzed (Participants) | 14 | 5 | 5
days
  Baseline hospitalization | 54 [20.0 to 63.5] | NA [NA to NA] — No patient hospitalized at start of RW-phase | NA [NA to NA] — No patient hospitalized at start of RW-phase
  Subsequent hospitalization | 5.5 [4.0 to 32.0] | 0 [0 to 0] | 0 [0 to 0]

17. Secondary Outcome: Change in Physician Global Assessment (PGA)
Description: The PGA is a direct surrogate of how a patient functions and assesses the severity of disease-related (auto-inflammatory) symptoms by selecting an integer score from 0 (no impact on subject; no symptoms) to 10 (no normal activities possible; highest severity of symptoms possible).
  The outcome lists the change from baseline of treatment phase to end of treatment phase/study in the PGA symptom severity score.
Time Frame: 34 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Single Arm Open-Label - Tadekinig Alfa | Randomized Withdrawal - Tadekinig Alfa Arm | Randomized Withdrawal - Placebo Arm
Number analyzed (Participants) | 14 | 5 | 5
score | -5.8 (2.1) | 0.4 (0.89) | 2.0 (3.39)

18. Secondary Outcome: Change in Patient/Caregiver Qualitative Evaluation of Health Status in Randomized Withdrawal Phase
Description: The individual disease-related symptoms score is the sum of (x) individual symptom scores within domain each ranging from 0 (None) to 5 (Very severe) for: general wellbeing (5), gastrointestinal (7), musculoskeletal (5), skin (2), eye (2), central nervous system (3), and lymphatic (2). Highest values indicate more severe disease-related symptoms within total score range from 0-130.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Randomized Withdrawal - Tadekinig Alfa Arm | Randomized Withdrawal - Placebo Arm
Number analyzed (Participants) | 3 | 2
score
  Start of RW phase | 11.3 (8.6) | 2.0 (2.8)
  End of RW phase | 7.7 (7.1) | 46.0 (14.1)
  Change from start to end of RW phase | -3.7 (5.7) | 44.0 (17.0)

19. Secondary Outcome: Immunogenicity Evaluation
Description: Generation of anti-recombinant human IL-18BP (anti-rhIL-18BP) antibodies
Time Frame: 34 weeks (SAOL + RW phases)
Reporting Status: Not Posted, anticipated posting 2026-03

20. Secondary Outcome: Local Tolerability at the Injection Site (as Defined by Number of Participants With Adverse Events of Special Interest)
Description: Adverse events of special interest (AESIs) are defined for this protocol as injection site reactions (including pruritus, erythema, swelling).
Time Frame: 34 weeks (SAOL + RW phases)
Population: Patients reporting at least one AESI. The safety and efficacy analyses during the SAOL phase is based on the SAOL-FAS as defined in the study protocol and statistical analysis plan. 1 patient treated with Placebo in the first treatment phase under the initial protocol design starting with a randomized treatment phase is excluded from the efficacy analysis due to the difference in treatment schedule but included in the safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Open-Label - Tadekinig Alfa | Randomized Withdrawal - Tadekinig Alfa Arm | Randomized Withdrawal - Placebo Arm
Number analyzed (Participants) | 14 | 5 | 5
Participants | 8 | 3 | 1

21. Secondary Outcome: Disease Reactivation Rate
Description: Disease reactivation rate for individual subjects (number of disease reactivations experienced per week while each subject is on the study treatment during the SAOL phase)
Time Frame: 18 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Disease reactivation rate per week
Arm/Group | Single Arm Open-Label - Tadekinig Alfa
Number analyzed (Participants) | 14
Disease reactivation rate per week | 0.0 (0.09)

22. Secondary Outcome: Treatment Failures
Description: Treatment failures (i.e. patients who experience at least one disease reactivation) during the SAOL phase
Time Frame: 18 weeks
Population: Treatment failures were defined as patients who experienced at least 1 disease reactivation. Disease reactivation includes full or partial disease reactivation after the first assessment indicating partial or complete response during the SAOL phase as defined in the statistical analysis plan.
  The safety and efficacy analyses during the SAOL phase is based on the SAOL-FAS as defined in the study protocol and statistical analysis plan.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Open-Label - Tadekinig Alfa
Number analyzed (Participants) | 14
Participants | 3

23. Other Pre Specified Outcome: Response to Therapy - Key Secondary Efficacy Endpoint
Description: Response to therapy (including complete response and partial response) in the SAOL phase from Week 10 onwards and observed at least at 2 consecutive visits at least 2 weeks apart during the SAOL phase
Time Frame: 18 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Open-Label - Tadekinig Alfa
Number analyzed (Participants) | 14
Participants | 10

ADVERSE EVENTS:
Time Frame: Adverse events were monitored and recorded for up to 34 weeks (from informed consent signature until completion of the study).
Description: Day to day fluctuations of the underlying disease of interest or other pre-existing disease or conditions present or detected at the start of the study were not to be reported as separate adverse events but assessed via the modified autoinflammatory disease index (mAIDAI) at scheduled or unscheduled visits in case of a disease reactivation.
Groups:
- Randomized Double-Blind Placebo-Controlled - Placebo Arm: The Randomized Double-Blind Placebo-Controlled (RDBPC) Analysis Set includes 1 patient treated with Placebo in the first treatment phase.
- Screening Phase: Time from informed consent signature up to day prior to first dose of study treatment
Arm/Group | Single Arm Open-Label - Tadekinig Alfa | Randomized Double-Blind Placebo-Controlled - Placebo Arm | Randomized Withdrawal - Tadekinig Alfa Arm | Randomized Withdrawal - Placebo Arm | Screening Phase
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/1 | 0/5 | 0/5 | 0/15
Serious Adverse Events (participants affected / at risk) | 3/14 | 0/1 | 0/5 | 0/5 | 1/15
Other Adverse Events (participants affected / at risk) | 14/14 | 1/1 | 4/5 | 4/5 | 7/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Open-Label - Tadekinig Alfa (N=14) | Randomized Double-Blind Placebo-Controlled - Placebo Arm (N=1) | Randomized Withdrawal - Tadekinig Alfa Arm (N=5) | Randomized Withdrawal - Placebo Arm (N=5) | Screening Phase (N=15)
Pyrexia (General disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Open-Label - Tadekinig Alfa (N=14) | Randomized Double-Blind Placebo-Controlled - Placebo Arm (N=1) | Randomized Withdrawal - Tadekinig Alfa Arm (N=5) | Randomized Withdrawal - Placebo Arm (N=5) | Screening Phase (N=15)
Injection site bruising (General disorders) | 5 (41) | 0 (0) | 2 (9) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 4 (10) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 4 (15) | 0 (0) | 2 (5) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (10) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Condition aggravated (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 2 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Secretion discharge (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 4 (6) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Red blood cell sedimentation rate increased (Investigations) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Adenovirus test positive (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Coronavirus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Human rhinovirus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interleukin-2 receptor increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sapovirus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum ferritin increased (Investigations) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vital signs measurement (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (5) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery dilatation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fontanelle bulging (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hypertension (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inflammatory bowel disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Food poisoning
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Teething (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatosplenomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (10) | 0 (0) | 0 (0) | 1 (8) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronavirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epstein-Barr viraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
External ear cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-09-03): https://cdn.clinicaltrials.gov/large-docs/60/NCT03113760/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/60/NCT03113760/SAP_001.pdf